CLINICAL TRIAL: NCT01936870
Title: DRUG USE INVESTIGATION FOR TOVIAZ
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0221096
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-01

CONDITIONS: Overactive Bladder (OAB)
Keywords: Toviaz; Fesoterodine; Post marketing surveillance; Japanese; Overactive Bladder; OAB; Good post marketing practice; Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fesoterodine (Toviaz)
  Interventions: Drug: Fesoterodine (Toviaz)

INTERVENTIONS:
Drug: Fesoterodine (Toviaz) — Fesoterodine 4 mg or 8 mg orally. Toviaz will be dosed according to labeling. The administration and duration of therapy will be determined by the treating physician to meet the patient's needs for treatment.

SUMMARY:
The purpose of this study is to collect effectiveness and safety information of fesoterodine related to their appropriate use in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed fesoterodine (Toviaz).

Exclusion Criteria:

* There are no exclustion criteria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prescribed fesoterodine (Toviaz) by investigators involved in protocol A0221096.
Sampling Method: Probability Sample
Enrollment: 2521 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221096&StudyName=Drug%20Use%20Investigation%20for%20Toviaz%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine Fumarate: Participants received fesoterodine fumarate at an oral dose of 4 mg once daily. The dose was increased up to 8 mg once daily according to symptoms.
Period: Overall Study
Arm/Group | Fesoterodine Fumarate
Started | 2492
Completed | 2303
Not Completed | 189
Not completed — No Visit After Treatment | 176
Not completed — Protocol Violation | 12
Not completed — No Drug Administration | 1

BASELINE CHARACTERISTICS:
Population: A total of 2492 participants completed this study. Of the 2492 participants, 189 participants were excluded from the baseline analysis due to following reasons: no visit after treatment (176 participants), protocol violation (12 participants), and no drug administration (1 participant).
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2303
Age, Customized [Count of Participants; unit: Participants]
  <15 years | 1
  >=15 and <65 years | 529
  ˃=65 years | 1773
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1228
  Male | 1075

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to fesoterodine fumarate in a participant who received fesoterodine fumarate. Relatedness to fesoterodine fumarate was assessed by the investigator.
Time Frame: 12 Weeks
Population: The safety analysis set comprised of participants who had satisfied the inclusion criteria of the study, and who had received fesoterodine fumarate at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2303
Participants | 415

2. Primary Outcome: Clinical Efficacy Rate
Description: Clinical efficacy rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Overall effectiveness of fesoterodine fumarate was determined by the investigator based on clinical symptoms and examinations. Clinical effectiveness was assessed according to the following categories: (1) effective, (2) ineffective, or (3) unassessable at week 12 of the treatment.
Time Frame: 12 Weeks
Population: The effectiveness analysis set comprised of subjects from the safety analysis set who had effectiveness evaluation at least once after treatment with fesoterodine fumarate, excluding those with off-label use.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2300
Percentage of participants | 74.8 [73.0 to 76.5]

3. Secondary Outcome: Number of Participants With Treatment-Related Serious Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to fesoterodine fumarate in a participant who received fesoterodine fumarate. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to fesoterodine fumarate was assessed by the investigator.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2303
Participants | 8

4. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to fesoterodine fumarate in a participant who received fesoterodine fumarate. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to fesoterodine fumarate was assessed by the investigator.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2303
Participants | 27

5. Secondary Outcome: Number of Participants With Adverse Events Related to Cognitive Function Disorder
Description: An adverse event was any untoward medical occurrence in a participant who received fesoterodine fumarate without regard to possibility of causal relationship. Adverse events related to cognitive function disorder were identified by broad searches on the Standard MedDRA Queries (SMQ).
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2303
Participants | 2

6. Secondary Outcome: Change From Baseline in the Mini-Mental State Examination (MMSE) Score at 12 Weeks
Description: Mini-Mental State Examination (MMSE) measured general cognitive functioning: orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons. Total score derived from sub-scores; total ranged from 0 to 30, higher score indicates better cognitive state. Mean change from baseline in the MMSE score at 12 weeks was presented along with the corresponding standard deviation.
Time Frame: Baseline, 12 Weeks
Population: The safety analysis set comprised of participants who had satisfied the inclusion criteria of the study, and who had received fesoterodine fumarate at least once. Participants with observed change in MMSE score were included in table.
Measure: Mean (Standard Deviation); unit: Scale
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 56
Scale | 0.4 (1.29)

7. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Among Whom Received Concomitant CYP3A4 Inhibitors
Description: Cytochrome P450 3A4 (CYP3A4) inhibitors included atazanavir, clarithromycin, indinavir, itraconazole, nelfinavir, ritonavir, saquinavir, and telithromycin.
Time Frame: 12 Weeks
Population: The safety analysis set comprised of participants who had satisfied the inclusion criteria of the study, and who had received fesoterodine fumarate at least once. "Number Analyzed" signifies those participants who were evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2303
Participants
  Received Concomitant CYP3A4 Inhibitors: number analyzed (Participants) | 21
  Received Concomitant CYP3A4 Inhibitors | 6
  Not Received Concomitant CYP3A4 Inhibitors: number analyzed (Participants) | 2282
  Not Received Concomitant CYP3A4 Inhibitors | 409

8. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Among Whom Received Concomitant CYP2D6 Inhibitors
Description: Cytochrome P450 2D6 (CYP2D6) inhibitors included quinidine and paroxetine. A treatment-related adverse event was any untoward medical occurrence attributed to fesoterodine fumarate in a participant who received fesoterodine fumarate. Relatedness to fesoterodine fumarate was assessed by the investigator.
Time Frame: 12 Weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2303
Participants
  Received Concomitant CYP2D6 Inhibitors: number analyzed (Participants) | 65
  Received Concomitant CYP2D6 Inhibitors | 11
  Not Received Concomitant CYP2D6 Inhibitors: number analyzed (Participants) | 2238
  Not Received Concomitant CYP2D6 Inhibitors | 404

9. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Among Whose Dose Was Increased From 4 mg to 8 mg
Description: as for outcome 1
Time Frame: 12 Weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2303
Participants
  From 4 mg to 8 mg: number analyzed (Participants) | 181
  From 4 mg to 8 mg | 53
  4 mg: number analyzed (Participants) | 1989
  4 mg | 330
  8 mg: number analyzed (Participants) | 133
  8 mg | 32

10. Secondary Outcome: Satisfaction Rate
Description: Satisfaction rate, which was defined as the percentage of participants who were satisfied by fesoterodine fumarate treatment over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Satisfaction scale was assessed by the participants according to the following categories: (1) satisfied, (2) unsatisfied, (3) uncertain, or (4) unconfirmed.
Time Frame: 12 Weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 2300
Percentage of participants | 59.0 [57.0 to 61.0]

11. Secondary Outcome: Change From Baseline in the Overactive Bladder Symptom Score (OABSS) at 12 Weeks
Description: Overactive Bladder Symptom Score (OABSS) was defined as the sum score (0 to 15) of the following four OAB symptoms: daytime frequency (2 at maximum), nighttime frequency (3 at maximum), urgency (5 at maximum), and urgency incontinence (5 at maximum). Higher score indicates worse symptoms. Mean change from baseline in the OABSS at 12 weeks was presented along with the corresponding standard deviation.
Time Frame: Baseline, 12 Weeks
Population: The effectiveness analysis set comprised of participants from the safety analysis set who had effectiveness evaluation at least once after treatment with fesoterodine fumarate, excluding those with off-label use. Participants with observed change in OABSS were included in table.
Measure: Mean (Standard Deviation); unit: Scale
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 1389
Scale | -3.4 (3.04)

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine Fumarate
Serious Adverse Events (participants affected / at risk) | 12/2303
Other Adverse Events (participants affected / at risk) | 361/2303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine Fumarate (N=2303)
Pneumonia (Infections and infestations) | 1
Loss of consciousness (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Acute abdomen (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Urinary retention (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Condition aggravated (General disorders) | 1
Residual urine volume increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine Fumarate (N=2303)
Dry mouth (Gastrointestinal disorders) | 36
Constipation (Gastrointestinal disorders) | 72
Urinary retention (Renal and urinary disorders) | 24
Dysuria (Renal and urinary disorders) | 63
Thirst (General disorders) | 166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.